CLINICAL TRIAL: NCT03004521
Title: A Randomised Pragmatic Trial Comparing the Clinical and Cost Effectiveness of Lithium and Quetiapine Augmentation in Treatment Resistant Depression
Brief Title: Lithium Versus Quetiapine in Treatment Resistant Depression
Acronym: LQD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: University of Oxford (Other); Newcastle University (Other); Oxford Health NHS Foundation Trust (Other Government); Northumberland, Tyne and Wear NHS Foundation Trust (Other); South London and Maudsley NHS Foundation Trust (Other); Tees, Esk and Wear Valleys NHS Foundation Trust (Unknown); Sussex Partnership NHS Foundation Trust (Other); Avon and Wiltshire Mental Health Partnership NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTA 14/222/02
Record Dates: First submitted 2016-11-17; First posted 2016-12-29 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Lithium; Quetiapine; Augmentation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Quetiapine Fumarate; Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium (Active Comparator): Lithium will be prescribed to patients in this arm as an augmenter on top of a patient's existing antidepressant treatment.
  Interventions: Drug: Lithium
- Quetiapine (Experimental): Quetiapine will be prescribed to patients in this arm as an augmenter on top of a patient's existing antidepressant treatment.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — Quetipatine prescribed in addition to the patient's existing antidepressant treatment.
  Arms: Quetiapine
Drug: Lithium — Lithium prescribed in addition to the patient's existing antidepressant treatment.
  Arms: Lithium

SUMMARY:
LQD is a multicentre randomised clinical trial comparing the clinical and cost effectiveness of lithium versus quetiapine when used as add-on therapies to antidepressant medication for patients with treatment resistant depression. The Lithium versus Quetiapine in Depression (LQD) study will assess patients over 12 months to establish which (if any) treatment is more likely to improve TRD over a long duration of time. Professor Anthony Cleare is the Chief Investigator and recruitment began in November 2016.

DETAILED DESCRIPTION:
This 12 month parallel group, multi-centre, patient randomised, pragmatic, open label trial is comparing the clinical and cost-effectiveness of the decision to prescribe lithium versus quetiapine add-on treatment to antidepressant medication. There will be two parallel groups: 1) Quetiapine add-on to existing antidepressant medication; 2) Lithium add-on to existing antidepressant medication. 276 patients will be randomised 1:1 at baseline to the decision to prescribe either lithium or quetiapine, and treatment will then be undertaken by clinicians on a real world basis. All patients, regardless of their treatment status, will be followed up in the trial for one year. This is a superiority design whereby we hypothesise that quetiapine will be superior to lithium in terms of time to treatment discontinuation and average symptom burden (QIDS-SR) over 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Under the care of a GP and/or adult mental health services
2. Current episode of depression meeting DSM-5 criteria for major depressive disorder (MDD) - single or recurrent episode 3.17-item HAM-D score ≥ 14 - this cut-off reflects a pragmatic minimum severity of depression as also chosen in comparable studies such as STAR*D (Rush et al 2006, Trivedi et al 2006)

4.Any gender and aged 18 years or over 5.Meet criteria for treatment resistant depression (Fekadu et al., 2009a; Cleare et al., 2015): current episode has not responded to at least two antidepressants given for at least 6 weeks at minimum therapeutic dose defined as fluoxetine ≥20mg/day, paroxetine ≥20mg/day, sertraline ≥50mg/day, citalopram ≥20mg/day, escitalopram ≥10mg/day, venlafaxine ≥75mg/day, duloxetine ≥60 mg/day, mirtazapine ≥15mg/day, tricyclic antidepressant ≥125mg/day, and dosage as guided by the national Maudsley Prescribing Guidelines or BNF for any other antidepressant. Please note, relapse whilst on an antidepressant also counts as a failed treatment trial 6.Current antidepressant treatment has remained unchanged and at, or above, a therapeutic dose for ≥6 weeks 7.Provision of written, informed consent.

Exclusion Criteria:

1. Diagnosis of bipolar disorder (defined as meeting DSM-5 criteria for bipolar 1 or bipolar 2) on the MINI 7.0 (as recommended treatments are different for bipolar depression)
2. Diagnosis of current psychosis (as recommended treatments are different for current psychosis - antidepressants plus antipsychotics is the first-line treatment recommendation (NiCE, 2009; Cleare et al., 2015)
3. Adequate use of lithium or quetiapine during the current episode. An adequate dose of lithium is defined as the patient taking lithium for at least 4 weeks at an adequate dose (leading to a documented plasma concentration of >0.4mmol/L) and for quetiapine, prescription in the range of 150-300mg/d for 4 weeks or longer. Or, if the patient has taken an inadequate dose of lithium or quetiapine in the current episode, the patient and clinician are not willing to re-prescribe/take the medication.
4. Ongoing use of another atypical antipsychotic (discontinuation will be required before study entry i.e. any time prior to randomisation)
5. Known contraindication to use of either lithium or quetiapine: known hypersensitivity of lithium or quetiapine or any of their excipients; severe renal insufficiency / impairment; untreated hypothyroidism; severe cardiac disease / insufficiency; low sodium levels e.g. dehydrated patients or those on low sodium diets; Addison's disease; Brugada syndrome or family history of Brugada syndrome; the rare hereditary inborn errors of metabolism galactosaemia, the Lapp lactase deficiency or glucose-galactose malabsorption; concomitant administration of cytochrome P450 3A4 inhibitors; or congenital QT prolongation.
6. We will not recruit any individual who is currently participating in a clinical trial of an investigational medical product (CTIMP).
7. Insufficient degree of comprehension or attention to be able to engage in trial procedures.
8. We will exclude women who are pregnant, actively trying for pregnancy, or currently breastfeeding. This will be based on verbal report of the subject. Otherwise the management will be as appropriate according to standard clinical practice within the context of a pragmatic, open trial, for example adequate contraceptive precautions decided on the clinical judgement of the prescriber.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Longitudinal depressive symptom severity | 52 weeks
  QIDS-SR
Difference in time to all-cause treatment discontinuation | 12 months
  The difference in the time at which patients stop taking the medication for any reason between the two treatment arms.

SECONDARY OUTCOMES:
Change in clinician rated depression severity | From baseline to weeks 8 and 52
  MADRS
Response rates | 8 weeks and 52 weeks
  Assessed using the MADRS questionnaire
Remission rates | 8 and 52 weeks
  Assessed using the MADRS questionnaire
Health related quality of life | Measured at 8 and 52 weeks
  Assessed using the EuroQol-5D questionnaire
Social functioning | Measured at baseline, 8 and 52 weeks
  Measured using the WSAS self rated questionnaire
Adherence to treatment | Measured at weeks 8 and 52
  Assessed using the MARS-5 questionnaire
Change in weight in kilograms | Measured at 8 and 52 weeks
  Assessed by weighing participants
Change in diastolic blood pressure | Change from baseline to 8 and 52 weeks
  Assessed by measuring blood pressure
Change in systolic blood pressure | Change from baseline to 8 and 52 weeks
  Assessed by measuring blood pressure
Time to uptake of a new intervention (pharmacological or non-pharmalogical) | 12 months
  Assessed by recording all pharmacological and non-pharmacological interventions
Time to initiation of treatment | Up to 12 months
  Assessed using treatment initiation form
CGI Global Improvement | Measured at 8 and 52 weeks
  CGI
Side effects | Measured at 8 and 52 weeks
  PRISE total score
Serious Adverse Events | 52 weeks
  Serious adverse events will be monitored and reported throughout the patient's participation in the trial.

OTHER OUTCOMES:
Change in global severity | Measured at 8, 26 and 52 weeks
  Change in CGI severity score
Global efficacy | Measured at 8, 26 and 52 weeks
  Change in CGI efficacy score
Side effects | Measured at 8 and 52 weeks
  Frequency of individual items on the PRISE
Physical health changes | Measured at baseline, 8, 26 and 52 weeks
  Not completed for all participants. Will be reported if there is a sufficient number e.g. blood parameters and waist circumference
Satisfaction with lithium / quetiapine treatment | Measured at 8, 26 and 52 weeks
  Measured using TSQM subscales
Change in self-report manic symptoms | Measured at baseline, 8, 26 and 52 weeks
  Measured using the Altman Mania Self Rating Scale
Change in anxiety symptoms | Measured at baseline, 8, 26 and 52 weeks
  GAD-7 score
Time to prescription | 0-52 weeks
  First date participant is given a prescription for the treatment
Baseline adherence to antidepressant | Measured at baseline
  MARS-5 score
Change in cognition | Measured at baseline, 8, 26 and 52 weeks
  Total DSCT score
Adherence of clinicians | 0-52 weeks
  Clinician adherence to prescribing and monitoring guidelines
Proportion of participants having an adequate treatment trial | 0-8 weeks
  Adequate treatment trial as defined in study protocol
Number of hospital admissions for depressive episode | 52 weeks
  Measured using psychiatric history assessment
Change in personality measure | Measured at baseline, 8, 26 and 52 weeks
  SAPAS
Social functioning | Measured weekly over 12 months
  WSAS
Economic analysis | 52 weeks
  Costs from the NHS and Personal Social Services perspective and from a societal perspective.
Predictors of treatment response | 52 weeks
  Measured using the Maudsley Staging Model, HAM-D, MINI 7, IDS-C and SAPAS questionnaires.
Longitudinal depression severity until time to all cause treatment discontinuation | 52 weeks
  Measured weekly using the QIDS-SR
Collection and analysis of biological samples for genetic, cytokine and cortisol analysis | 0-52 weeks
  Blood/hair/saliva samples collected in collaboration with the BRC BioResource
Reliability and validity of the Maudsley VAS | Measured at baseline, 8, 26 and 52 weeks
  Measured using the Maudsley VAS, validated against the QIDS-SR and MADRS
Discrepancy between the self-rated and clinician-rated version of 16 item IDS | Measured at baseline and 8 weeks
  Assessed using QIDS and IDS
Relationship between quetiapine and lithium serum levels, prescribed dose and depressive symptom severity | 52 weeks
  MADRS
Time to new interventions for depression. | 52 weeks
  Measured using concomitant medication and concomitant therapy questionnaires
Number of new interventions for depression | 52 weeks
  Measured using concomitant medication and concomitant therapy questionnaires
Patient rated experience of the True Colours weekly monitoring system | 8 / 26 / 52 weeks
  Qualitative Interview in a subset of participants
Change in cognitive function | Baseline, 8, 26 and 52 weeks
  THINC-it composite and individual tests scores in a subset of participants
12. Patient views and experiences of lithium and quetiapine | 52 week visit
  Qualitative interviews in a subset of participants

CONTACTS AND LOCATIONS:
Overall Officials: Anothony Cleare, Principal Investigator — Professor of Psychiatry
Locations (1):
- Institute of Psychiatry, Psychology and Neuroscience, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The decision to share IPD to other researchers will be made by the CI on a case by case basis.

REFERENCES:
- [Derived] Marwood L, Taylor R, Goldsmith K, Romeo R, Holland R, Pickles A, Hutchinson J, Dietch D, Cipriani A, Nair R, Attenburrow MJ, Young AH, Geddes J, McAllister-Williams RH, Cleare AJ. Study protocol for a randomised pragmatic trial comparing the clinical and cost effectiveness of lithium and quetiapine augmentation in treatment resistant depression (the LQD study). BMC Psychiatry. 2017 Jun 26;17(1):231. doi: 10.1186/s12888-017-1393-0. PMID 28651526
- See also: Study website link — https://www.kcl.ac.uk/research/lqd-study